CLINICAL TRIAL: NCT04770012
Title: Early Initiation of Antiplatelet ThERapy In HeArt TranspLantation: AERIAL Trial
Brief Title: AERIAL Trial: Antiplatelet Therapy in Heart Transplantation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-version 1.0
Record Dates: First submitted 2021-01-25; First posted 2021-02-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Allograft Vasculopathy; Heart Transplant
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: 2:2:1 randomization to placebo-control, aspirin 81 mg daily or clopidogrel 75 mg daily
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, clinical care providers and research staff will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel
- aspirin (Active Comparator)
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: Placebo — patients randomized to placebo study group will be dispensed placebo capsules to be taken daily for the duration of the treatment
  Arms: placebo
Drug: aspirin — patients randomized to aspirin study group will be dispensed aspirin capsules to be taken daily for the duration of the treatment
  Arms: aspirin
Drug: Clopidogrel — patients randomized to clopidogrel study group will be dispensed clopidogrel capsules to be taken daily for the duration of the treatment
  Other Names: plavix
  Arms: clopidogrel

SUMMARY:
Cardiac allograft vasculopathy is a common complication affecting heart transplant patients. This condition causes narrowing of the heart arteries leading to graft dysfunction. The research team is investigating whether early antiplatelet therapy post heart transplant can prevent the development of CAV. This study will determine the feasibility of a large multicenter randomized placebo-controlled trial to answer this question.

DETAILED DESCRIPTION:
Heart transplant patients who fulfill selection criteria will undergo baseline clinical evaluation and data collection. Participants will be randomized to either placebo, aspirin or clopidogrel to be taken daily for the duration of the study. Patients will undergo invasive coronary studies (angiography, optical coherence tomography and intracoronary flow) and platelet function testing at 2 and 12 months post heart transplant. In addition, angiography will be performed at 24 months post heart transplant and thereafter according to institutional protocol. The primary analysis will determine the feasibility of conducting a large multicenter randomized placebo controlled trial by assessing recruitment rates, event rates, treatment crossovers and loss to follow-up. Secondary analyses will include assessing the effect of antiplatelet treatment on angiographic CAV, coronary intimal disease on optical coherence tomography, coronary macrovascular and microvascular function by intracoronary flow measures, and platelet function.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant
2. Age ≥18 years
3. Able to provide informed consent

Exclusion Criteria:

1. Allergy or known intolerance to aspirin
2. Allergy or known intolerance to clopidogrel
3. Intracranial hemorrhage ≤14 days
4. Bleeding disorder
5. Platelet count <50 x 109/L
6. History of aspirin related gastrointestinal bleeding or ulcers
7. Non-cardiac indication for antiplatelet therapy
8. Anticoagulation >3 months
9. Allergy to iodinated contrast
10. Unable to undergo coronary angiography due to glomerular filtration rate ≤30 mL/min/1.73 m2 for non-dialysis patients
11. Unable to undergo coronary angiography due to unsuitable vascular access
12. Combined solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment rate | 3 years
  Average recruitment rate of 4.5 patients per month at 3 study sites
Feasibility: CAV event rate | 3 years
  2-year CAV event rate of >8%
Feasibility: Treatment cross over rate | 3 years
  Crossover from aspirin to placebo <2%, clopidogrel to placebo <2%, placebo to aspirin <4%, placebo to clopidogrel <1%
Feasibility: Loss to follow up rate | 3 years
  Loss-to-follow-up <1%
Feasibility: Compliance to treatment | 3 years
  Compliance to treatment >80%

SECONDARY OUTCOMES:
Cardiac allograft vasculopathy | 1 and 2 years post transplant
  Angiographic CAV disease severity according to ISHLT CAV 0-3 grading
Coronary intimal disease | 2 months, 1 year post transplant
  Coronary intimal volume measured on OCT
Coronary endothelial function | 2 months and 1 year post transplant
  Coronary flow reserve measured by intracoronary flow assessment
Coronary macrovascular function | 2 months and 1 year post transplant
  Fractional flow reserve measured by intracoronary flow assessment
Coronary microvascular function | 2 months and 1 year post transplant
  Index of microcirculatory resistance measured by intracoronary flow assessment
Platelet Function | Baseline, 2 months and 1 year post transplant
  Assessment of response to antiplatelet therapy using Enzyme-Linked Immunosorbent Assays (ELISA) for thromboxane B2 and Vasodilator Stimulated Phosphoprotein (VASP).

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chih, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (3):
- Canada (3):
  - St.Pauls Hospital, Vancouver, British Columbia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital UHN, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rheaume M, Aleksova N, Madsen JC, Benichou G. Chronic Rejection Series: Heart Cardiac Allograft Vasculopathy. Transplantation. 2026 Jan 1;110(1):e28-e41. doi: 10.1097/TP.0000000000005453. Epub 2025 Jul 14. PMID 40653611